CLINICAL TRIAL: NCT05016843
Title: The Study of Internet-delivered, Transdiagnostic Treatments for Anxiety and Depression ("TRAnsdiagnostisk BEhandling (Elektronisk)")
Brief Title: The Study of Internet-delivered, Transdiagnostic Treatments for Anxiety and Depression
Acronym: TRAbee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stockholm University (Other)
Responsible Party: Principal Investigator, Per Carlbring, Professor, Stockholm University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: TRAbee
Record Dates: First submitted 2021-08-08; First posted 2021-08-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Anxiety Disorders; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- CBT, 8 weeks and access to forum. (Experimental)
  Interventions: Behavioral: Treatment condition: Internet-administered Unified protocol; Other: Treatment length: 8 weeks; Other: Access to a moderated forum
- CBT, 16 weeks and access to forum. (Experimental)
  Interventions: Behavioral: Treatment condition: Internet-administered Unified protocol; Other: Treatment length: 16 weeks; Other: No access to a moderated forum
- CBT, 8 weeks and no access to forum. (Experimental)
  Interventions: Behavioral: Treatment condition: Internet-administered Unified protocol; Other: Treatment length: 8 weeks; Other: No access to a moderated forum
- CBT, 16 weeks and no access to forum. (Experimental)
  Interventions: Behavioral: Treatment condition: Internet-administered Unified protocol; Other: Treatment length: 16 weeks; Other: Access to a moderated forum
- Psychodynamic therapy, 8 weeks and access to forum. (Experimental)
  Interventions: Behavioral: Treatment condition: Internet-administered Affect phobia treatment; Other: Treatment length: 8 weeks; Other: Access to a moderated forum
- Psychodynamic therapy, 16 weeks and access to forum. (Experimental)
  Interventions: Behavioral: Treatment condition: Internet-administered Affect phobia treatment; Other: Treatment length: 16 weeks; Other: Access to a moderated forum
- Psychodynamic therapy, 8 weeks and no access to forum. (Experimental)
  Interventions: Behavioral: Treatment condition: Internet-administered Affect phobia treatment; Other: Treatment length: 8 weeks; Other: No access to a moderated forum
- Psychodynamic therapy, 16 weeks and no access to forum. (Experimental)
  Interventions: Behavioral: Treatment condition: Internet-administered Affect phobia treatment; Other: Treatment length: 16 weeks; Other: No access to a moderated forum
- Waitlist, 8 weeks and access to forum. (Experimental)
  Interventions: Other: Treatment condition: Waitlist control; Other: Treatment length: 8 weeks; Other: Access to a moderated forum
- Waitlist, 16 weeks and access to forum. (Experimental)
  Interventions: Other: Treatment condition: Waitlist control; Other: Treatment length: 16 weeks; Other: Access to a moderated forum
- Waitlist, 8 weeks and no access to forum. (Experimental)
  Interventions: Other: Treatment condition: Waitlist control; Other: Treatment length: 8 weeks; Other: No access to a moderated forum
- Waitlist, 16 weeks and no access to forum. (Experimental)
  Interventions: Other: Treatment condition: Waitlist control; Other: Treatment length: 16 weeks; Other: No access to a moderated forum

INTERVENTIONS:
Behavioral: Treatment condition: Internet-administered Unified protocol — Treatment condition:
  The cognitive, behavioral treatment Unified protocol is a transdiagnostic treatment for anxiety and depression. Participants are taught five techniques in order to find new and more helpful ways to react to hindering thoughts and feelings: mindfulness, cognitive flexibility, identify and reduce behavioral avoidance, increase willingness to experience physiological sensations and exposure. The intervention is delivered online through a secure platform. Modules consist of text and the participants can work with the material whenever they wish to. Participants gain access to a new treatment modul every week.
  Arms: CBT, 16 weeks and access to forum.; CBT, 16 weeks and no access to forum.; CBT, 8 weeks and access to forum.; CBT, 8 weeks and no access to forum.
Behavioral: Treatment condition: Internet-administered Affect phobia treatment — The aim of psychodynamic Affect phobia treatment is for the patient to reach an intellectual and emotional understanding of his/hers problems. The goal of the treatment is for participants to decrease emotional avoidance and start to approach emotions and increase emotional awareness. Participants are taught this through linking their symptoms to their emotional avoidance, observe frequent and maladaptive patterns in relationships and see how these are linked to emotional avoidance. The intervention is delivered online through a secure platform. Modules consist of text and the participants can work with the material whenever they wish to. Participants gain access to a new treatment modul every week.
  Arms: Psychodynamic therapy, 16 weeks and access to forum.; Psychodynamic therapy, 16 weeks and no access to forum.; Psychodynamic therapy, 8 weeks and access to forum.; Psychodynamic therapy, 8 weeks and no access to forum.
Other: Treatment condition: Waitlist control — The waitlist condition is a control condition without any intervention.
  Arms: Waitlist, 16 weeks and access to forum.; Waitlist, 16 weeks and no access to forum.; Waitlist, 8 weeks and access to forum.; Waitlist, 8 weeks and no access to forum.
Other: Treatment length: 8 weeks — Participants will partake in their treatment condition for 8 weeks.
  Arms: CBT, 8 weeks and access to forum.; CBT, 8 weeks and no access to forum.; Psychodynamic therapy, 8 weeks and access to forum.; Psychodynamic therapy, 8 weeks and no access to forum.; Waitlist, 8 weeks and access to forum.; Waitlist, 8 weeks and no access to forum.
Other: Treatment length: 16 weeks — Participants will partake in their treatment condition for 16 weeks.
  Arms: CBT, 16 weeks and access to forum.; CBT, 16 weeks and no access to forum.; Psychodynamic therapy, 16 weeks and access to forum.; Psychodynamic therapy, 16 weeks and no access to forum.; Waitlist, 16 weeks and access to forum.; Waitlist, 16 weeks and no access to forum.
Other: Access to a moderated forum — During their treatment, participants will have access to a discussion forum moderated by a clinician. Participants are encouraged to discuss questions and experiences related to their treatment condition.
  Arms: CBT, 16 weeks and no access to forum.; CBT, 8 weeks and access to forum.; Psychodynamic therapy, 16 weeks and access to forum.; Psychodynamic therapy, 8 weeks and access to forum.; Waitlist, 16 weeks and access to forum.; Waitlist, 8 weeks and access to forum.
Other: No access to a moderated forum — Participants will not have access to a moderated forum, hence their treatment is self-guided.
  Arms: CBT, 16 weeks and access to forum.; CBT, 8 weeks and no access to forum.; Psychodynamic therapy, 16 weeks and no access to forum.; Psychodynamic therapy, 8 weeks and no access to forum.; Waitlist, 16 weeks and no access to forum.; Waitlist, 8 weeks and no access to forum.

SUMMARY:
Anxiety and depression are common psychiatric disorders, resulting in suffering and impaired functioning for the individual. Today, most psychological treatments are disorder specific, even tough comorbidity between depression and anxiety and different anxiety disorders is rule rather than exception. Transdiagnostic treatments target the common features between depression and anxiety disorders and has shown to be as effective as disorder specific treatments in reducing symptoms of the disorders. Unified protocol and Affect phobia treatment are two types of transdiagnostic treatments that, to our knowledge, never been compared in research before. Internet-administered treatment presents a promising way to increase availability of psychotherapeutic interventions such as transdiagnostic treatments. However, questions regarding the optimal treatment length and level of support remain unanswered. The aim of this study is to examine two internet-administered transdiagnostic treatments and their effect on anxiety and depression, and to investigate the impact of treatment length and access to a moderated forum.

The study will investigate three factors: type of transdiagnostic treatment, length of treatment and whether patients have access to a moderated forum or not. 2400 participants with anxiety and/or depression will be randomly assigned to one of 12 subgroups and subsequently offered treatment based on differing combinations of the previously mentioned factors (200 participants/arm). The treatment conditions are internet-administered cognitive, behavioral treatment (CBT) Unified protocol and the psychodynamic Affect phobia treatment as well as a waitlist control group. Participants will also be randomized to either 8 or 16 weeks of treatment and access to a moderated forum or not.

Primary outcome measures will be the Patient Health Questionnaire, the Generalized Anxiety Disorder 7-item scale and the Brief Quality of Life scale. Negative effects of treatment will also be assessed. In addition to pre- and post-treatment measurements, the study includes one mid-treatment and three follow-up assessments (6, 12 and 24 months).

ELIGIBILITY:
Inclusion Criteria:

* Be able to read and write Swedish,
* access to a mobile phone/computer,
* 18 years or older,
* GAD-7 ≥ 5 and/or
* PHQ-9 ≥ 10.

Exclusion Criteria:

* Partaking in other psychological treatment,
* has started or adjusted treatment with psychopharmacological drugs for anxiety, worry or depression within the nearest month,
* severe depression (PHQ-9 ≥ 20) or suicidal (PHQ-9, item 9>2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2477 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2026-01-22 (Actual); Study Completion 2026-01-22 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9-item scale (PHQ-9) | Through study completion, an average of 2 years.
  The PHQ-9 features nine items for assessing depression in a clinical context and screening of depression in the general population.
Generalised Anxiety Disorder 7- item scale (GAD-7) | Through study completion, an average of 2 years.
  The GAD-7 features seven items for assessing anxiety and screening for generalized anxiety disorder.
Brunnsviken Brief Quality of Life Scale (BBQ) | Through study completion, an average of 2 years.
  The BBQ features 12 items concerning 6 areas of life rated on importance and satisfaction.

SECONDARY OUTCOMES:
The Personality Inventory for DSM Short Form (PID-5) | Baseline only.
  The PID-5 is a self-rated measure of personality-related problems featuring 25 items.
Negative Effects Questionnaire (NEQ) | At post-treatment only (which is week 8 or 16 depending on treatment allocation).
  The NEQ measures unwanted effects of treatments.
Reflective Functioning Questionnaire 8 (RFQ-8) | Through study completion, an average of 2 years.
  RFQ features 8 items assessing the ability to understand mental states of the self and others.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Derived] Hlynsson JI, Carlbring P. Diagnostic accuracy and clinical utility of the PHQ-2 and GAD-2: a comparison with long-format measures for depression and anxiety. Front Psychol. 2024 May 10;15:1259997. doi: 10.3389/fpsyg.2024.1259997. eCollection 2024. PMID 38800678
- [Derived] Hlynsson JI, Lindner P, Barri B, Carlbring P. Exploring cutoff points and measurement invariance of the Brunnsviken brief quality of life inventory. Front Psychol. 2024 Jan 8;14:1305682. doi: 10.3389/fpsyg.2023.1305682. eCollection 2023. PMID 38259555